CLINICAL TRIAL: NCT05514080
Title: A Pilot Study to Evaluate Eli Lilly's Insulin Dosing Algorithm to Control Glycemia in Insulin-treated Adults With Type 2 Diabetes
Brief Title: A Study to Evaluate Eli Lilly's Insulin Dosing Algorithm to Control Glycemia in Insulin-treated Adults With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-5837
Record Dates: First submitted 2020-12-01; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Insulin pump therapy; Eli Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Insulin alone closed-loop (Other)
  Interventions: Other: Insulin closed-loop

INTERVENTIONS:
Other: Insulin closed-loop — 41-hour intervention period in which the participants are treated with rapid insulin in the closed-loop system.

SUMMARY:
The objective of this study is to generate preliminary data in an inpatient setting to help optimize an insulin dosing logic (that decides how much to deliver insulin) for Eli Lilly's system.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants giving written informed consent will undergo an admission visit to determine eligibility for study entry. Participants who meet the inclusion and exclusion criteria will then participate in two 41-hour intervention visits using Eli Lilly's insulin dosing algorithm.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, all participants must meet the following criteria:

1. Adult male or female ≥ 18 years of age.
2. Type 2 diabetes mellitus has been clinically diagnosed (the diagnosis of type 2 diabetes is based on the investigator's judgment) for at least 12 months
3. Using multiple daily insulin injections (one basal and ≥ 2 prandial doses) for ≥ 3 months.
4. Using insulin glargine (U100 or U300), detemir, degludec, or NPH.
5. Most recent (in the last 6 month) HbA1c ≤ 10%.
6. Use of a GLP1 agonist or SGLT inhibitor for the past 3 months.

Exclusion Criteria:

Participants who meet any of the following criteria are not eligible for the study:

1. Severe hypoglycaemic episode ≤ two months before admission.
2. Ongoing pregnancy, or any newly diagnosed pregnancy throughout the study
3. Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
4. Recent (within the past 6 months) acute macrovascular event (e.g. acute coronary syndrome or cardiac surgery).
5. Peripheral vascular disease, foot ulcer, Charcot arthropathy or any condition that limits ability to walk
6. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
7. Use of oral hypoglycaemic agents besides SGLTi's, GLP1 agonists, and or metformin and unwilling to discontinue for the run-in and intervention period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Glucose outcomes: percentage of time spent in specific glucose ranges (ex: 3.9-10.0 mmol/L) | 24 hours
  As this is a pilot study, the only primary outcome is the glucose outcomes during the closed-loop portion.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tsoukas, MD, Principal Investigator — Royal Victoria Hospital, Belfast
Locations (1):
- Centre for Innovative Medicine at McGill University Health Centre Research Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Effect of intensive blood-glucose control with metformin on complications in overweight patients with type 2 diabetes (UKPDS 34). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):854-65. PMID 9742977
- [Background] Nathan DM, Buse JB, Davidson MB, Ferrannini E, Holman RR, Sherwin R, Zinman B; American Diabetes Association; European Association for the Study of Diabetes. Medical management of hyperglycaemia in type 2 diabetes mellitus: a consensus algorithm for the initiation and adjustment of therapy: a consensus statement from the American Diabetes Association and the European Association for the Study of Diabetes. Diabetologia. 2009 Jan;52(1):17-30. doi: 10.1007/s00125-008-1157-y. Epub 2008 Oct 22. PMID 18941734
- [Background] Riddle MC, Rosenstock J, Gerich J; Insulin Glargine 4002 Study Investigators. The treat-to-target trial: randomized addition of glargine or human NPH insulin to oral therapy of type 2 diabetic patients. Diabetes Care. 2003 Nov;26(11):3080-6. doi: 10.2337/diacare.26.11.3080. PMID 14578243
- [Background] Pickup JC, Keen H, Parsons JA, Alberti KG. Continuous subcutaneous insulin infusion: an approach to achieving normoglycaemia. Br Med J. 1978 Jan 28;1(6107):204-7. doi: 10.1136/bmj.1.6107.204. PMID 340000
- [Background] Reznik Y, Cohen O, Aronson R, Conget I, Runzis S, Castaneda J, Lee SW; OpT2mise Study Group. Insulin pump treatment compared with multiple daily injections for treatment of type 2 diabetes (OpT2mise): a randomised open-label controlled trial. Lancet. 2014 Oct 4;384(9950):1265-72. doi: 10.1016/S0140-6736(14)61037-0. Epub 2014 Jul 2. PMID 24998009
- [Background] Thabit H, Tauschmann M, Allen JM, Leelarathna L, Hartnell S, Wilinska ME, Acerini CL, Dellweg S, Benesch C, Heinemann L, Mader JK, Holzer M, Kojzar H, Exall J, Yong J, Pichierri J, Barnard KD, Kollman C, Cheng P, Hindmarsh PC, Campbell FM, Arnolds S, Pieber TR, Evans ML, Dunger DB, Hovorka R. Home Use of an Artificial Beta Cell in Type 1 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2129-2140. doi: 10.1056/NEJMoa1509351. Epub 2015 Sep 17. PMID 26379095
- [Background] Haidar A, Legault L, Matteau-Pelletier L, Messier V, Dallaire M, Ladouceur M, Rabasa-Lhoret R. Outpatient overnight glucose control with dual-hormone artificial pancreas, single-hormone artificial pancreas, or conventional insulin pump therapy in children and adolescents with type 1 diabetes: an open-label, randomised controlled trial. Lancet Diabetes Endocrinol. 2015 Aug;3(8):595-604. doi: 10.1016/S2213-8587(15)00141-2. Epub 2015 Jun 8. PMID 26066705
- [Background] Haidar A, Rabasa-Lhoret R, Legault L, Lovblom LE, Rakheja R, Messier V, D'Aoust E, Falappa CM, Justice T, Orszag A, Tschirhart H, Dallaire M, Ladouceur M, Perkins BA. Single- and Dual-Hormone Artificial Pancreas for Overnight Glucose Control in Type 1 Diabetes. J Clin Endocrinol Metab. 2016 Jan;101(1):214-23. doi: 10.1210/jc.2015-3003. Epub 2015 Nov 2. PMID 26523526
- [Background] Gingras V, Rabasa-Lhoret R, Messier V, Ladouceur M, Legault L, Haidar A. Efficacy of dual-hormone artificial pancreas to alleviate the carbohydrate-counting burden of type 1 diabetes: A randomized crossover trial. Diabetes Metab. 2016 Feb;42(1):47-54. doi: 10.1016/j.diabet.2015.05.001. Epub 2015 Jun 10. PMID 26072052
- [Background] Taleb N, Emami A, Suppere C, Messier V, Legault L, Ladouceur M, Chiasson JL, Haidar A, Rabasa-Lhoret R. Efficacy of single-hormone and dual-hormone artificial pancreas during continuous and interval exercise in adult patients with type 1 diabetes: randomised controlled crossover trial. Diabetologia. 2016 Dec;59(12):2561-2571. doi: 10.1007/s00125-016-4107-0. Epub 2016 Oct 4. PMID 27704167
- [Background] Haidar A, Messier V, Legault L, Ladouceur M, Rabasa-Lhoret R. Outpatient 60-hour day-and-night glucose control with dual-hormone artificial pancreas, single-hormone artificial pancreas, or sensor-augmented pump therapy in adults with type 1 diabetes: An open-label, randomised, crossover, controlled trial. Diabetes Obes Metab. 2017 May;19(5):713-720. doi: 10.1111/dom.12880. Epub 2017 Mar 8. PMID 28094472
- [Background] Gingras V, Haidar A, Messier V, Legault L, Ladouceur M, Rabasa-Lhoret R. A Simplified Semiquantitative Meal Bolus Strategy Combined with Single- and Dual-Hormone Closed-Loop Delivery in Patients with Type 1 Diabetes: A Pilot Study. Diabetes Technol Ther. 2016 Aug;18(8):464-71. doi: 10.1089/dia.2016.0043. Epub 2016 May 18. PMID 27191385